CLINICAL TRIAL: NCT04124601
Title: Neoadjuvant CHemoradiotherapy With Sequential Ipilimumab and NivOlumab in RECtal Cancer (CHINOREC): a Prospective Randomized, Open-label, Multicenter, Phase II Clinical Trial
Brief Title: Neoadjuvant Chemoradiotherapy With Sequential Ipilimumab and Nivolumab in Rectal Cancer
Acronym: CHINOREC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Laengle, MD, PhD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Johannes Laengle, MD, PhD, Sponsor-Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-7HJ; 2019-003865-17 (EudraCT Number)
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Rectal Cancer
Keywords: Ipilimumab; Nivolumab; Chemoradiotherapy; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Neoadjuvant Chemoradiotherapy (Other): Neoadjuvant Chemoradiotherapy (50 Gy in 2 Gy fractions + Capecitabine 1650 mg/m2/d over 25 working days)
  Interventions: Radiation: Chemoradiotherapy
- Neoadjuvant Chemoradiotherapy, Ipilimumab, Nivolumab (Experimental): Neoadjuvant Chemoradiotherapy (50 Gy in 2 Gy fractions + Capecitabine 1650 mg/m2/d over 25 working days) with sequential Ipilimumab (1 mg/kg IV on day 7) and Nivolumab (3 mg/kg IV on day 14, 28 and 42)
  Interventions: Radiation: Chemoradiotherapy; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Radiation: Chemoradiotherapy — Capecitabine tablet with fractionated radiotherapy
  Other Names: Radiochemotherapy; Chemoradiation
Drug: Ipilimumab — Infusion
  Other Names: Yervoy®
  Arms: Neoadjuvant Chemoradiotherapy, Ipilimumab, Nivolumab
Drug: Nivolumab — Infusion
  Other Names: Opdivo®
  Arms: Neoadjuvant Chemoradiotherapy, Ipilimumab, Nivolumab

SUMMARY:
This prospective randomized, open-label, multicenter, phase II clinical trial investigates the safety and tolerability of standard neoadjuvant chemoradiotherapy (CRT) with sequential ipilimumab and nivolumab in rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* All sexes
* Histologically confirmed carcinoma of the rectum
* Suitable for local therapy with curative intent
* Medical need for a standard neoadjuvant CRT
* Suitable to withstand a course of standard neoadjuvant CRT
* Written informed consent form (ICF) for participation in the study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Metastatic disease that is considered incurable by local therapies
* Previous surgery of the tumor other than biopsy
* Pregnancy, breastfeeding or expectancy to conceive
* Disagreement of participants with reproductive potential to use contraception throughout the study period and for up to 180 days after the last dose of study therapy
* Prior therapy with anti-CTLA-4, anti-PD-1, anti-PD-L1, anti-PD-L2 or any other agent directed against co-inhibitory T cell receptors or has previously participated in clinical studies with immunotherapy
* Any contraindication according to the official medical information of Ipilimumab or Nivolumab
* Live vaccine within 30 days prior to the first dose of study therapy
* Hepatitis B or C
* Human immunodeficiency virus (HIV)
* Immunodeficiency
* Allogeneic tissue or solid organ transplantation
* Autoimmune disease that has required systemic therapy in the past 2 years with modifying agents, steroids or immunosuppressive drugs
* Systemic steroids or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Active non-infectious pneumonitis
* Active infection requiring systemic therapy
* Treatment with botanical preparations (i.e. herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to randomization/treatment
* Participants with serious or uncontrolled medical disorders
* Uncontrolled or significant cardiovascular disease (myocardial infarction, uncontrolled angina, any history of clinically significant arrhythmias, QTc prolongation in males > 450 ms and > 470 ms in females, participants with history of myocarditis)
* Allergies and adverse drug reaction (history of allergy or hypersensitivity to study drug components, contraindications to any of the study drugs of the chemotherapy regimen)
* Other exclusion criteria: Prisoners or participants who are involuntarily incarcerated, participants who are compulsorily detained for treatment of either a psychiatric or physical (i.e. infectious disease) illness
* White blood cells < 2000/μL (SI: < 2.00 × 109/L)
* Neutrophils < 1500/μL (SI: < 1.50 × 109/L)
* Platelets < 100 × 103/μL (SI: < 100 × 109/L) (transfusions not permitted within 72 h prior to qualifying laboratory value)
* Hemoglobin < 9.0 g/dl (SI: < 90 g/L) (transfusions not permitted within 72 h prior to qualifying laboratory value)
* Serum creatinine > 1.5 × upper limit of normal (ULN) or calculated creatinine clearance < 50 ml/min (using the Cockcroft-Gault formula)
* AST/ALT: > 3.0 × ULN
* Total bilirubin > 1.5 × ULN (except participants with Gilbert Syndrome who must have a total bilirubin level of < 3.0 × ULN)
* Troponin T (TnT) or I (TnI) > 2 × institutional ULN. TnT or TnI levels between > 1 to 2 × ULN will be permitted to participate in the study if a repeat assessment remains 2 × ULN and participant undergoes a cardiac evaluation. When repeat levels within 24 h are not available, a repeat test should be conducted as soon as possible.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | 20 weeks
  Incidence of treatment-emergent adverse events will be assessed according to the latest "Clavien- Dindo Classification of surgical complications" and Common Terminology Criteria of Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Radiographic therapy response between pre-and post-neoadjuvant treatment | 20 weeks
  Radiographic therapy response will be determined by magnetic resonance imaging-assessed tumor regression grade (mrTRG)
Pathologic therapy response to neoadjuvant treatment | 20 weeks
  Pathological therapy response will be determined according to the latest American Joint Committee on Cancer/International Union Against Cancer-Tumor Node Metastasis (AJCC/UICC-TNM) staging and tumor regression grade (TRG).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bergmann, MD, Principal Investigator — Division of Visceral Surgery, Department of General Surgery, Medical University of Vienna
Locations (5):
- Austria (5):
  - State Hospital Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Congregational Hospital Linz - Sisters of Mercy, Linz
  - Hospital of St. John of God, Vienna
  - Medical University of Vienna, Vienna
  - Hospital North - Clinic Floridsdorf, Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laengle J, Kuehrer I, Kulu A, Kabiljo J, Ammon D, Zirnbauer R, Stift A, Herbst F, Dauser B, Monschein M, Razek P, Haegele S, Biebl M, Geinitz H, Hulla W, Kalinina P, Mullauer L, Widder J, Bittermann C, Pils D, Tamandl D, Laengle F, Schmid R, Bergmann M. Dual Immune Checkpoint Inhibition Plus Neoadjuvant Chemoradiotherapy in Rectal Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2527769. doi: 10.1001/jamanetworkopen.2025.27769. PMID 40844778